CLINICAL TRIAL: NCT01910389
Title: Phosphodiesterase Type 5 Inhibition With Tadalafil Changes Outcomes in Heart Failure
Acronym: PITCH-HF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated by funding agency
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01HL105463 (NIH)
Record Dates: First submitted 2013-07-25; First posted 2013-07-29 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2014-01

CONDITIONS: Heart Failure; Pulmonary Hypertension
Keywords: Heart failure; Pulmonary hypertension; tadalafil; Phosphodiesterase Type 5 Inhibition
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tadalafil (Active Comparator): Tadalafil is supplied in 20 mg tablets. Subjects will take 20 mg (one tablet) once per day and will be titrated to 40 mg (two tablets once per day) after one week. Subjects are on study drug for the duration of the trial.
  Interventions: Drug: Tadalafil
- Placebo (Placebo Comparator): Placebo of tadalafil. Subjects will take one tablet once per day and will be titrated to two tablets once per day after one week. Subjects are on study drug for the duration of the trial.
  Interventions: Drug: Placebo for tadalafil

INTERVENTIONS:
Drug: Tadalafil
  Other Names: Adcirca
  Arms: Tadalafil
Drug: Placebo for tadalafil
  Arms: Placebo

SUMMARY:
This study is a multi-center, prospective, randomized, double blind, placebo-controlled clinical trial. Subjects in the study will be adults with New York Heart Association (NYHA) Class II-IV heart failure (HF) due to left ventricular systolic dysfunction (LVSD), left ventricular ejection fraction (LVEF) <0.40, and secondary pulmonary hypertension (PH). The purpose of the study is to evaluate the safety, effectiveness, and effects of tadalafil compared to placebo on the subjects' functional capacity / quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 21 years or older.
* NYHA Class II-IV HF with LVSD (most recent LVEF < 0.40).
* At high risk of future clinical instability, indicated by EITHER:

a hospitalization for the primary reason of decompensated HF within the 12 months prior to screening; OR a plasma B-type Natriuretic Peptide (BNP) level ≥ 300 pg/ml or N-terminal prohormone of brain natriuretic peptide (NT-proBNP) ≥1800pg/ml measured during a period of clinical stability in the 3 months prior to screening.

* Documented secondary PH within the last 6 months
* Medication and device treatment according to current American Heart Association/American College of Cardiology (AHA/ACC) guidelines.
* Stable medical therapy for 30 days prior to randomization
* African-American patients intolerant of or otherwise unable or unwilling to utilize isosorbide dinitrate/hydralazine therapy will be included.
* Willingness to comply with protocol, attend follow-up appointments, complete all study assessments and provide written informed consent.

Exclusion Criteria:

* Concurrent or anticipated nitrate use for any reason, or nitrate use within the 14 days prior to screening through the day of randomization.
* Known allergy, hypersensitivity (anaphylaxis), or adverse reaction to tadalafil or other Phosphodiesterase Type 5 (PDE5) inhibitor
* Erectile dysfunction treated with a PDE5 inhibitor.
* Severe renal dysfunction defined as an estimated glomerular filtration rate (GFR) < 30 ml/min/1.73 m^2 or requiring chronic dialysis
* Current use of alpha antagonists (except carvedilol or tamsulosin) or use of cytochrome P450 3A4 inhibitors (ketoconazole, itraconazole, erythromycin, or cimetidine). Patients who have used a protease inhibitor that is a P450 3A4 inhibitor for longer than one week can be enrolled.
* Pulmonary arterial hypertension (World Health Organization (WHO) Group I, III-V) for which PDE5 inhibitor therapy may be indicated
* Severe pulmonary disease requiring home oxygen therapy
* Comorbidities including clinically significant valvular stenosis (aortic valve area < 0.8 cm^2 or a mitral valve area <1.0 cm^2), uncontrolled hypertension (systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg) or hypotension (systolic blood pressure <85 mmHg)
* Chronic intravenous inotrope therapy
* Non-arteritic anterior ischemic optic neuropathy (NAION)
* ST elevation MI (STEMI) within 90 days prior to screening
* Coronary Artery Bypass Grafting (CABG) or mitral valve surgery, initiation of cardiac resynchronization (CRT) or initiation of β-blocker therapy within the 6 months prior to screening
* Infiltrative or inflammatory myocardial disease (e.g. amyloid, sarcoid)
* Heart transplant recipient
* United Network Organ Sharing (UNOS) status 1A or 1B
* Mechanical circulatory support (MCS) use or planned MCS use at time of consent
* Active malignancy (except non-melanoma skin cancer) requiring therapy other than observation.
* Severe non-cardiac illness resulting in life expectancy judged less than three years
* Known chronic hepatic disease defined as aspartate aminotransferase (AST) and alanine transaminase (ALT) levels > 3.0 times the upper limit of normal
* Inability to walk even a few steps due to non-cardiac (e.g. orthopedic) reasons
* Participation in any clinical trial within the last 30 days (with exception of observational study)
* Previous randomization in PITCH-HF

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc J. Semigran, MD, Principal Investigator — Massachusetts General Hospital; Susan F Assmann, PhD, Principal Investigator — New England Research Institutes, Inc.; Flora S Siami, MPH, Principal Investigator — New England Research Institutes, Inc.
Locations (63):
- United States (62):
  - Heart Center Inc - Research, Huntsville, Alabama
  - Baptist Health Transplant Institute, Little Rock, Arkansas
  - Allianz Medical and Research Center, Fountain Valley, California
  - Christiana Care Health System, Newark, Delaware
  - Broward Health, Fort Lauderdale, Florida
  - Miller School of Medicine University of Miami, Miami, Florida
  - Orlando Health, Orlando, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Brevard Cardiovascular Research Associates, Rockledge, Florida
  - University Cardiology Associates LLC, Augusta, Georgia
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Illinois Hospital, Chicago, Illinois
  - Methodist Medical Group Cardiology, Peoria, Illinois
  - Baptist Hospital East, Louisville, Kentucky
  - Research Integrity LLC, Owensboro, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Primary Care Cardiology Research, Inc., Ayer, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - MGH West, Waltham, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Covenant Center for the Heart, Saginaw, Michigan
  - Essentia Health East, Duluth, Minnesota
  - Metropolitan Heart and Vascular Institute, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Missouri Cardiovascular Specialists, Columbia, Missouri
  - St. Luke's Health System, Kansas City, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Heart & Vascular Center of NJ/Cardio Metabolic Institute, Somerset, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Columbia University Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Cardiology Associates of Schenectady, Schenectady, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Bronx - Lebanon Hospital Center, The Bronx, New York
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - The Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Dayton VA Medical Center, Dayton, Ohio
  - Oklahoma City VA, Oklahoma City, Oklahoma
  - Warren Cancer Research Foundation, Tulsa, Oklahoma
  - Lancaster Heart and Stroke Foundation, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Grand View - Lehigh Valley Health Service, Sellersville, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - CIVA/CArdiovascular Research Institute of Dallas, Dallas, Texas
  - Michael E. Debakey VA Medical Center, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Aspirus Wausau Hospital, Wausau, Wisconsin
- Jewish General Hospital, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tadalafil | Placebo
Started | 15 | 8
Completed | 0 | 0
Not Completed | 15 | 8
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Study Closed | 13 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil | Placebo | Total
Number analyzed (Participants) | 15 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 4 | 14
  >=65 years | 5 | 4 | 9
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.6 [42.3 to 72.5] | 63.3 [51.7 to 76.8] | 62.6 [47.7 to 73.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 13 | 7 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 14 | 8 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 11 | 6 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Composite Outcome of Cardiovascular (CV) Mortality or Heart Failure (HF) Hospitalization
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 3 years per subject
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cardiovascular Mortality
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 3 years per subject
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Heart Failure Hospitalization
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 3 years per subject
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: All-cause Mortality
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 3 years per subject
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Composite Outcome of All-cause Mortality or CV Hospitalization (Myocardial Infarction, Acute Coronary Syndrome, Stroke, Arrhythmia, or Heart Failure)
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 3 years per subject
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Frequency of CV Hospitalizations
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 3 years per subject
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Frequency of HF Hospitalizations
Time Frame: Randomization through each subject's last semi-annual visit, up to a maximum of 3 years per subject
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in 6 Minute Walk Distance From Baseline to 3 Months
Time Frame: Randomization to 3 months
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in MLHFQ Score From Baseline to 3 Months
Time Frame: Randomization to 3 months
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in 6 Minute Walk Distance From Baseline to 18 Months
Time Frame: Randomization to 18 months
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Trend in 6 Minute Walk Distance From Baseline Through 18 Months
Time Frame: Randomization to 18 months
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) Score From Baseline to 18 Months
Time Frame: Randomization to 18 months
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Trend in Minnesota Living With Heart Failure Questionnaire (MLHFQ) Score From Baseline Through 18 Months
Time Frame: Randomization to 18 months
Population: Trial was terminated early. Data for outcome not obtained.
Arm/Group | Tadalafil | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include any untoward medical occurrence which occurred after a subject gave informed consent and no later than 30 days after a subject permanently discontinued the study medication, for a maximum of 3 years per subject
Description: If a subject experiences more than 1 of a given AE within a system organ class (SOC), the subject was counted only once for that AE.
Arm/Group | Tadalafil | Placebo
Serious Adverse Events (participants affected / at risk) | 4/15 | 2/8
Other Adverse Events (participants affected / at risk) | 3/15 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=15) | Placebo (N=8)
CHF EXACERBATION (Cardiac disorders) | 0 (0) | 1 (2)
CHF EXACERBATION, DYSPNEA (Cardiac disorders) | 0 (0) | 1 (1)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
HOSPITALIZATION FOR DECOMPENSATED HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0)
ER ADMISSION; NOSEBLEED (General disorders) | 1 (1) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil (N=15) | Placebo (N=8)
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0)
FLUSHING (Vascular disorders) | 1 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 0 (0)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (2) | 0 (0)
METALLIC TASTE TO FOOD (General disorders) | 1 (2) | 0 (0)
PALPITATIONS (Cardiac disorders) | 1 (1) | 0 (0)
STOMACH UPSET (Gastrointestinal disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects. Outcome measure data not obtained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes